CLINICAL TRIAL: NCT04376619
Title: Alert Kidney Intervention
Brief Title: Preventing Acute Kidney Injury
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: never was able to recruit
Sponsor: Atlantic Health System (Other)
Responsible Party: Principal Investigator, Shivangi K. Patel, Principal Investigator, Atlantic Health System
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 1527104-1
Record Dates: First submitted 2020-04-27; First posted 2020-05-06 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Intervention Model Description: Two part study: all patients will be triaged by alert system whether they are high risk for acute kidney injury and those patients that are identified as high risk for AKI have standard of care implemented by following kidney disease improving global outcomes guidelines in preventing AKI and part 2 will perform procedure called remote ischemic preconditioning in addition to standard of care in part1 in those patients that are identified as high risk for acute kidney injury.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KDIGO guidelines (Experimental): Part 1 of study, those identified as high risk for AKI then will have Kidney Disease Global Improving outcomes guideline implemented to see if this reduces incidence of AKI
  Interventions: Other: KDIGO guidelines
- RIPC (Experimental): part 2 of study, those identified as high risk of AKI will have Kidney Disease Improving Global Outcomes guidelines and RIPC implemented to see if this reduces incidence of AKI compared to part 2 of study
  Interventions: Other: remote ischemic preconditioning

INTERVENTIONS:
Other: remote ischemic preconditioning — inflation and deflation of cuff 5min each cycle repeated 3 times
  Arms: RIPC
Other: KDIGO guidelines — KDIGO stands for Kidney disease Improving global outcomes guidelines, and have guidelines for prevention and treatment of AKI which is considered standard of care.
  Arms: KDIGO guidelines

SUMMARY:
Acute kidney injury increases the risk for chronic kidney disease, length of stay, readmissions and mortality. Currently the only way to diagnose acute kidney injury is with a serum creatinine or drop in urine output. Biomarkers for acute kidney injury are well elevated before rise in creatinine. Hypothesis is that by implementing an electronic alert system with an algorithm followed by remote ischemic preconditioning will prevent acute kidney injury.

DETAILED DESCRIPTION:
The propose study is to incorporate an alert system in current medical health system and an algorithm will be used to activate clinicians and Nephrologist to confirm if patient is at high risk. Once identified as high risk the clinician and/or nephrologist will intervene and change current management if needed. First phase of study will look at an alert system and algorithm was enough to lower incidence of acute kidney injury. Phase 2 will also use alert system and algorithm that will be further randomized those that are identified as high risk for acute kidney injury to remote ischemic preconditioning.

ELIGIBILITY:
Inclusion Criteria:

* any admitted patients that are not excluded by exclusion criteria
* Patients who's creatinine returns to baseline after admitted can be included in study if patient still remains admitted.

Exclusion Criteria:

* End stage renal disease
* estimated glomerular filtration rate less then 20
* Left ventricular assist device patients
* observation status
* hospice patients
* pregnancy
* age less then 18
* acute kidney injury on admission defined as 1.5 times elevated creatinine prior to last admission's creatinine
* nephrology consult already placed
* renal transplant or nephrectomy within 1 year
* Patients unable to provide consent

exclusion for remote ischemic preconditioning in addition to above exclusion will be:

* symptoms or diagnosis of peripheral arterial disease
* Patients in shock defined by requiring inotropes or vasopressors

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
number of participants who developed acute kidney injury | during hospitalization, up to three months
  development of acute kidney injury as measured by serum creatinine 1.5 times more then baseline
number of participants who required dialysis | during hospitalization, up to three months
  need for initiation of dialysis after acute kidney injury develops during the admission

SECONDARY OUTCOMES:
number of participants who are placed on hospice or have expired | at time of admission when enrolled in study to 1 year post discharge
  death or placed on hospice
progression to chronic kidney disease | at time of admission when enrolled in study to 1 year post discharge
  measured by serum creatinine over 1 year on followup labs
number of participants who receive dialysis | at time of admission when enrolled in study to 1 year post discharge
  initiation of dialysis starting from at time of admission to 1 year post discharge
number of participants who are readmitted | discharged from when enrolled in study to 1 year post discharge
  readmissions to hospital within 1 year of first admission date
length of stay | during hospitalization, up to three months
  starting from onset of acute kidney injury measured by elevated creatinine 1.5 times baseline creatinine to last day of discharged

CONTACTS AND LOCATIONS:
Overall Officials: Shivangi Patel, M.D., Principal Investigator — atlantich health system

IPD SHARING:
Plan to Share IPD: Yes
excel file that is password protected, only to those involved in the study directly
Supporting Information: Study Protocol, SAP, ICF
Time Frame: six months at end of study and for 3 more months post study completion
Access Criteria: must be involved in implementing /executing the study